# Study protocol

Twenty years of pancreatic surgery in Iceland: a retrospective cohort study

### **Background:**

Pancreatic surgery is often occasioned by cancer in the pancreas or periampullary region, where pancreatic ductal adenocarcinoma (PDAC) is the most common diagnosis. This disease has a dire prognosis and is projected to soon surpass breast cancer as the third leading cause of cancer death in the European Union. The overall 5-year survival rate is reported to be 10% in the US, to a large extent due to the fact that 80-85% of patients are inoperable at diagnosis. Survival after resection is better but not high, reported to be between 20 and 25% 5 years after surgery. Periampullary tumors – including ampullary, duodenal and distal bile duct carcinomas – have a better survival with a postoperative 5-year survival rate of around 45%. Apart from these diagnoses, pancreatic surgery is occasionally performed due to neuroendocrine tumors, chronic pancreatitis, metastases from renal cancer, and, increasingly, for premalignant cystic lesions such as intraductal papillary mucinous neoplasms (IPMN). 3, 4

Pancreatic operations are large and complex procedures, with reported rates of severe complications (Clavien-Dindo ≥3a) after pancreaticoduodenectomy (PD) between 20 and 30% in modern data, and up to 38% after total pancreatectomy.<sup>5,6</sup> Distal pancreatectomy (DP) is a smaller procedure where the most usual postoperative complication is leakage of pancreatic fluid from the divided pancreas.<sup>7</sup> Minimally invasive pancreatic surgery has come the furthest among distal resections, where three randomized controlled trials have now shown the safety of the technique both from a perioperative and an oncological perspective.<sup>7-9</sup> Recent international guidelines recommend minimally invasive distal pancreatectomy (MIDP) to be considered for benign, pre-malignant and malignant lesions alike in the pancreatic body or tail.<sup>10</sup>

The question of volume in pancreatic surgery has been a growing topic over the last decade, with many studies indicating an advantage in terms of rate of resections, rate of radical resections, short-term and overall mortality with increasing hospital volume. <sup>11-13</sup> Current international recommendations for training in minimally invasive pancreatic resections recommend an annual hospital volume of 50 PDs and 10 DPs to qualify for a training program. <sup>14</sup>

Iceland is a small country in a unique situation, with a population of 380 000 people and situated on the border of the North Atlantic and Arctic oceans. <sup>15</sup> There is one university hospital in the capital of Reykjavik, performing the majority of the surgery and all of the malignancy surgery on the island. As this is by necessity a low-volume hospital in terms of pancreatic surgery, there is a long tradition of specialists training overseas to gain sufficient experience and volumes to be able to maintain a good standard of care despite the isolated

conditions of the island. There is, however, limited information available on the outcomes of pancreatic surgery in the country.

The aim of this study is to investigate the outcomes of pancreatic surgery in Iceland over the last 20 years.

## **Study characteristics:**

This is a retrospective cohort study with data accessed from patients' medical journals.

### **Patients:**

All patients who have undergone pancreatic resection in Iceland between 2002-2022 will be included in the study. For the secondary outcome of duodenal cancer, patients with duodenal cancer who did not undergo resection in the same time span will also be included.

## **Primary outcome:**

The primary outcome of the study is the rate of severe complications and short-term mortality after pancreatic resections in Iceland.

### **Secondary outcomes:**

- Demographic, operative and postoperative data after pancreatic resections compared between operation methods.
- Oncological data and survival among patients with pancreatic and periampullary cancer.
- Outcomes after pancreatic surgery among patients who underwent resection for cystic lesions.
- Comparison of patients who underwent minimally invasive distal pancreatectomy during the study period to those who underwent open distal resection.
- Demographic and histopathological data as well as survival compared between patients with duodenal cancer who underwent resection and patients who did not.
- Trends over time in the usage of pancreatic and minimally invasive surgery as well as changes in outcomes.

# Variables accessed from the medical journals of patients:

| Preoperative data | Operative data | Postoperative data | Histopathological data<br>and survival |
|---|---|---|---|
| Age | Operation date | Clavien-Dindo complication score <sup>16</sup> | TNM stage |
| Gender | Operation time | Postoperative pancreatic fistula <sup>17</sup> | Radicality |
| Body mass index | Type of operation | Delayed gastric emptying <sup>18</sup> | Lymph nodes acquired and positive |
| Comorbidities | Minimally invasive or open | Postpancreatectomy hemorrhage <sup>19</sup> | Histopathological diagnosis |
| Preoperative medicines including statins | Type of pancreatic anastomosis | Bile leak <sup>20</sup> | Oncologic treatment including details |
| ASA score | Blood loss | Postpancreatectomy acute pancreatitis <sup>21</sup> | Date of recurrence |
| ECOG performance status | Arterial or venous resection | Blood and drain<br>amylase and bilirubin<br>levels | Date of death |
| Unintended weight loss | Additional organ resection | Days with drain | |
| Smoking | Splenectomy | Radiologic drain placement | |
| Date of diagnosis | | Intensive care and days | |
| Date of treatment decision | | Reoperation and details | |
| Date of multidisciplinary conference | | Wound dehiscence | |
| Preoperative biliary drainage | | Wound infection | |
| Preoperative endoscopic ultrasound | | Pneumonia | |
| Other preoperative intervention | | Cardiovascular complications | |
| Preoperative blood tests:<br>CEA, Ca 19-9,<br>hemoglobin, bilirubin,<br>albumin | | Neurological complications | |
| Preoperative cyst fluid tests | | Thromboembolism | |
| Preoperative biopsy | | Length of hospital stay | |
| Preoperative TNM stage | | In-hospital mortality | |
| Preoperative assessment<br>(resectable, borderline,<br>locally advanced or<br>metastasized) | | Textbook outcome <sup>22</sup> | |
| Neoadjuvant<br>chemotherapy including<br>details | | | |

ASA, American Society of Anesthesiologists; ECOG, Eastern Cooperative Oncology Group; TNM, tumor, node, metastasis.

#### Time frame:

- Developing study protocol and seeking ethical permission: summer of 2023.
- Data collection: autumn of 2023 to spring of 2024.
- Data analyses and writing of manuscript: rest of 2024.
- Publication: 2025.

#### **References:**

- 1. Mizrahi JD, Surana R, Valle JW, Shroff RT. Pancreatic cancer. *Lancet*. 2020;**395**(10242):2008-20.
- 2. RCC. Pancreatic Cancer: National Practice Guidelines (in Swedish). Regionala cancercentrum i samverkan. 2021.
- 3. Tanaka M, Fernández-Del Castillo C, Kamisawa T, Jang JY, Levy P, Ohtsuka T, et al. Revisions of international consensus Fukuoka guidelines for the management of IPMN of the pancreas. *Pancreatology*. 2017;**17**(5):738-53.
- 4. European evidence-based guidelines on pancreatic cystic neoplasms. *Gut*. 2018;**67**(5):789-804.
- 5. Gleeson EM, Pitt HA, Mackay TM, Wellner UF, Williamsson C, Busch OR, et al. Failure to Rescue After Pancreatoduodenectomy: A Transatlantic Analysis. *Ann Surg*. 2021;**274**(3):459-66.
- 6. Latenstein AEJ, Mackay TM, Beane JD, Busch OR, van Dieren S, Gleeson EM, et al. The use and clinical outcome of total pancreatectomy in the United States, Germany, the Netherlands, and Sweden. *Surgery*. 2021;**170**(2):563-70.
- 7. de Rooij T, van Hilst J, van Santvoort H, Boerma D, van den Boezem P, Daams F, et al. Minimally Invasive Versus Open Distal Pancreatectomy (LEOPARD): A Multicenter Patient-blinded Randomized Controlled Trial. *Ann Surg.* 2019;**269**(1):2-9.
- 8. Björnsson B, Larsson AL, Hjalmarsson C, Gasslander T, Sandström P. Comparison of the duration of hospital stay after laparoscopic or open distal pancreatectomy: randomized controlled trial. *Br J Surg.* 2020;**107**(10):1281-8.
- 9. Korrel M, Jones LR, van Hilst J, Balzano G, Björnsson B, Boggi U, et al. Minimally invasive versus open distal pancreatectomy for resectable pancreatic cancer (DIPLOMA): an international randomised non-inferiority trial. *The Lancet Regional Health Europe*. 2023;**31**.
- 10. Abu Hilal M, van Ramshorst TME, Boggi U, Dokmak S, Edwin B, Keck T, et al. The Brescia Internationally Validated European Guidelines on Minimally Invasive Pancreatic Surgery (EGUMIPS). *Annals of Surgery*. 9900:10.1097/SLA.000000000000006006.
- 11. Lemmens VE, Bosscha K, van der Schelling G, Brenninkmeijer S, Coebergh JW, de Hingh IH. Improving outcome for patients with pancreatic cancer through centralization. *Br J Surg.* 2011;**98**(10):1455-62.
- 12. Gooiker GA, Lemmens VE, Besselink MG, Busch OR, Bonsing BA, Molenaar IQ, et al. Impact of centralization of pancreatic cancer surgery on resection rates and survival. *Br J Surg.* 2014;**101**(8):1000-5.
- 13. Onete VG, Besselink MG, Salsbach CM, Van Eijck CH, Busch OR, Gouma DJ, et al. Impact of centralization of pancreatoduodenectomy on reported radical resections rates in a nationwide pathology database. *HPB (Oxford)*. 2015;17(8):736-42.

- 14. Korrel M, Lof S, Alseidi AA, Asbun HJ, Boggi U, Hogg ME, et al. Framework for Training in Minimally Invasive Pancreatic Surgery: An International Delphi Consensus Study. *J Am Coll Surg*. 2022;**235**(3):383-90.
- 15. Icelandic population statistics, overview. *Statistics Iceland*. 2023 [Available from: <a href="https://www.statice.is/">https://www.statice.is/</a>.
- 16. Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. *Ann Surg.* 2004;**240**(2):205-13.
- 17. Bassi C, Marchegiani G, Dervenis C, Sarr M, Abu Hilal M, Adham M, et al. The 2016 update of the International Study Group (ISGPS) definition and grading of postoperative pancreatic fistula: 11 Years After. *Surgery*. 2017;**161**(3):584-91.
- 18. Wente MN, Bassi C, Dervenis C, Fingerhut A, Gouma DJ, Izbicki JR, et al. Delayed gastric emptying (DGE) after pancreatic surgery: a suggested definition by the International Study Group of Pancreatic Surgery (ISGPS). *Surgery*. 2007;**142**(5):761-8.
- 19. Wente MN, Veit JA, Bassi C, Dervenis C, Fingerhut A, Gouma DJ, et al. Postpancreatectomy hemorrhage (PPH): an International Study Group of Pancreatic Surgery (ISGPS) definition. *Surgery*. 2007;**142**(1):20-5.
- 20. Koch M, Garden OJ, Padbury R, Rahbari NN, Adam R, Capussotti L, et al. Bile leakage after hepatobiliary and pancreatic surgery: a definition and grading of severity by the International Study Group of Liver Surgery. Surgery. 2011;149(5):680-8.
- 21. Marchegiani G, Barreto SG, Bannone E, Sarr M, Vollmer CM, Connor S, et al. Postpancreatectomy Acute Pancreatitis (PPAP): Definition and Grading From the International Study Group for Pancreatic Surgery (ISGPS). *Ann Surg.* 2022;**275**(4):663-72.
- van Roessel S, Mackay TM, van Dieren S, van der Schelling GP, Nieuwenhuijs VB, Bosscha K, et al. Textbook Outcome: Nationwide Analysis of a Novel Quality Measure in Pancreatic Surgery. *Ann Surg.* 2020;**271**(1):155-62.